CLINICAL TRIAL: NCT03326193
Title: A Phase 2, Single-arm, Open-label Study to Evaluate the Safety and Efficacy of Niraparib Combined With Bevacizumab as Maintenance Treatment in Patients With Advanced Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer Following Front-line Platinum-based Chemotherapy With Bevacizumab
Brief Title: A Study of Niraparib Combined With Bevacizumab Maintenance Treatment in Participants With Advanced Ovarian Cancer Following Response on Front-Line Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213358; 3000-02-004 (Other: Tesaro)
Record Dates: First submitted 2017-10-10; First posted 2017-10-31 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Neoplasms
Keywords: Poly(adenosine diphosphate-ribose) polymerase (PARP) inhibitor; Ovarian Cancer; Primary Peritoneal carcinoma; Fallopian Tube; Vascular endothelial growth factor (VEGF) inhibitor; Bevacizumab; Niraparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Bevacizumab

STUDY DESIGN:
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving niraparib+ bevacizumab (Experimental): Participants will be administered bevacizumab 15 milligram per kilogram (mg/kg) via a 30 minute (min) intravenous (IV) infusion on Day 1 of each 21-day cycle. Niraparib will be administered orally once a day continuously throughout each 21-day cycle (84-day cycle after amendment 2). On Day 1 of each cycle, niraparib will be administered upon completion of bevacizumab infusion. The starting dose of niraparib will be based on the participant's Baseline actual body weight or platelet count.
  Interventions: Drug: Niraparib; Biological: Bevacizumab

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered orally once a day continuously throughout each 21 day cycle (84-day cycle after amendment 2). The starting dose of niraparib will be based on the participant's Baseline actual body weight or platelet count. Participants with a Baseline actual body weight of greater than equal to (>=) 77 kg and Baseline platelet count of >=150,000/ microliter (μL) will take 300 mg/day (3X100mg) at each dose administration. Participants with a Baseline actual body weight of less than (<) 77 kg and/or Baseline platelet count of <150,000/μL will take 200 mg (2X100 mg) at each dose administration.
  Other Names: ZEJULA
Biological: Bevacizumab — Maintenance bevacizumab 15 mg/kg will be administered via a 30-minute IV infusion on Day 1 of every 21-day cycle in the absence of progressive disease (PD), unacceptable toxicity, participant withdrawal, Investigator's decision, or death. Bevacizumab will be administered for up to 10 months during the maintenance phase or up to a total of 15 months inclusive of approximately 5 months of bevacizumab received with chemotherapy.
  Other Names: Avastin

SUMMARY:
Niraparib is an oral inhibitor of poly adenosine diphosphate-ribose polymerase (PARP)-1 and PARP-2. This study will evaluate safety and efficacy of niraparib combined with bevacizumab as maintenance treatment in participants with advanced (stage IIIB-IV) ovarian cancer, fallopian tube cancer, or primary peritoneal cancer following front-line platinum-based chemotherapy with bevacizumab. Eligible participants who achieve complete response (CR), partial response (PR), or no evidence of disease (NED) following treatment with platinum-based chemotherapy in addition to bevacizumab will be enrolled in the study and will receive maintenance treatment with niraparib (for up to 3 years) combined with bevacizumab (for up to 10 months during the maintenance phase or up to a total of 15 months inclusive of the approximately 5 months of bevacizumab received with chemotherapy) or until disease progression, unacceptable toxicity, participant withdrawal, Investigator's decision, or death, whichever comes first. Participants who have not progressed after 3 years of niraparib maintenance treatment may continue with niraparib beyond 3 years if they are benefiting from treatment, upon consultation with Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be female, be greater than equal to (>=) 18 years of age, be able to understand the study procedures, and agree to participate in the study by providing written informed consent.
* Participants must have newly diagnosed International Federation of Gynecology and Obstetrics (FIGO) Stage IIIB to IV epithelial ovarian, fallopian tube, or peritoneal cancer and have recovered from debulking surgery.
* Participants must have high-grade serous or endometrioid or high-grade predominantly serous or endometrioid histology, regardless of homologous recombination deficiency (HRD) or germline breast cancer susceptibility gene (gBRCA) mutation status. Participants with non mucinous epithelial ovarian cancer and gBRCA mutation are eligible.
* Participants must have completed front-line, platinum-based chemotherapy with CR, PR, or NED and have first study treatment dose within 12 weeks of the first day of the last cycle of chemotherapy:
* a. A platinum-based regimen must have consisted of a minimum of 6 and a maximum of 9 treatment cycles. Participants who discontinued platinum-based therapy early as a result of non hematologic toxicity specifically related to the platinum regimen (ie, neurotoxicity or hypersensitivity) are eligible if they have received a minimum of 4 cycles of the platinum regimen.
* b. IV, intraperitoneal, or neoadjuvant platinum-based chemotherapy is allowed; for weekly therapy, 3 weeks is considered 1 cycle. Interval debulking is allowed.
* Participants must have received, prior to enrollment, a minimum of 3 cycles of bevacizumab in combination with the last 3 cycles of platinum-based chemotherapy. Participants who undergo interval debulking surgery are eligible if they have received only 2 cycles of bevacizumab in combination with the last 3 cycles of platinum-based chemotherapy.
* Participant must have had 1 attempt at optimal debulking surgery.
* Participant must have either CA-125 in the normal range or CA-125 decrease by more than 90% during front-line therapy that is stable for at least 7 days (ie, no increase > 15% from nadir).
* Participant must have adequate organ function.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
* Participant must have normal blood pressure or well-controlled hypertension.
* Participant must agree to complete patient-reported outcome (PROs) (Functional Assessment of Cancer Therapy-Ovarian Symptom Index [FOSI] questionnaire) throughout the study, including after study treatment discontinuation.
* Participant must be able to take oral medication.
* Participant must agree to undergo tumor HRD testing at screening. The tumor sample must be confirmed to be available during the screening period and submitted after the participant has been enrolled. Participants do not have to wait for the HRD test result to be enrolled. If archival tumor tissue is not available for testing, the participant must agree to undergo a fresh biopsy.
* Participant of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin) within 72 hours prior to receiving the first dose of study treatment.
* Participants must be postmenopausal, free from menses for > 1 year, surgically sterilized, or willing to use adequate contraception to prevent pregnancy or must agree to abstain from activities that could result in pregnancy throughout the study, starting with enrollment through 180 days after the last dose of study treatment.

Exclusion Criteria:

* Participants with ovarian tumors of non-epithelial origin (eg, germ cell tumor) or any low grade tumors.
* Participants with clinically significant cardiovascular disease (eg, significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina < 6 months to enrollment, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade II or greater peripheral vascular disease, and history of cerebrovascular accident (CVA) within 6 months).
* Participants with gastrointestinal disorders or abnormalities that would interfere with absorption of study treatment.
* History of bowel obstruction, including sub-occlusive disease, related to the underlying disease or history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscesses. Evidence of rectosigmoid involvement by pelvic examination or bowel involvement on computed tomography (CT) scan or clinical symptoms of bowel obstruction.
* Participant has proteinuria as demonstrated by urine protein:creatinine ratio >= 1.0 at screening or urine dipstick for proteinuria ≥ 2 (participants discovered to have >=2 proteinuria on dipstick at baseline should undergo a 24-hour urine collection and must demonstrate < 2 gram (g) of protein in 24 hours to be eligible).
* Participant has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML).
* Participant has received treatment previously with a PARP inhibitor.
* Other than ovarian cancer, the participant has been diagnosed or treated for invasive cancer less than 5 years prior to study enrollment. Participants with cervical carcinoma in situ, non melanomatous skin cancer, and ductal carcinoma in situ definitively treated are allowed.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non malignant systemic disease, or active, uncontrolled infection.
* Participant has known contraindication to PARP inhibitors or (VEGF inhibitors.
* Participant is at increased bleeding risk due to concurrent conditions (eg, major injuries or surgery within the past 28 days prior to start of study treatment, history of CVA, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).
* Participant is immunocompromised (participants with splenectomy are allowed).
* Participant has known, active hepatic disease (ie, hepatitis B or C).
* Participant has a QT interval prolongation > 480 milliseconds (ms) at screening. If a participant has a prolonged QT interval and the prolongation is deemed to be due to a pacemaker upon Investigator evaluation (ie, the participant otherwise has no cardiac abnormalities), then the participant may be eligible to participate in the study following discussion with the Medical Monitor.
* Participant is pregnant, or expecting to conceive children while receiving study drug or for 180 days after the last dose of study drug ; additionally, female participant should not breastfeed during treatment with niraparib and for 30 days after receipt of the last dose due to the potential for serious adverse reactions from niraparib in breastfed infants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Englewood, New Jersey
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardesty MM, Krivak TC, Wright GS, Hamilton E, Fleming EL, Belotte J, Keeton EK, Wang P, Gupta D, Clements A, Gray HJ, Konecny GE, Moore RG, Richardson DL. OVARIO phase II trial of combination niraparib plus bevacizumab maintenance therapy in advanced ovarian cancer following first-line platinum-based chemotherapy with bevacizumab. Gynecol Oncol. 2022 Aug;166(2):219-229. doi: 10.1016/j.ygyno.2022.05.020. Epub 2022 Jun 9. PMID 35690498

RESULTS

PARTICIPANT FLOW:
Groups:
- Niraparib + Bevacizumab: Participants received bevacizumab 15 milligram per kilogram (mg/kg) via a 30 minute intravenous (IV) infusion on Day 1 of each 21-day cycle. Niraparib (200 mg or 300 mg) was administered orally once a day continuously throughout each 21-day cycle. On Day 1 of each 21-day cycle, niraparib was administered upon completion of bevacizumab infusion.
Period: Overall Study
Arm/Group | Niraparib + Bevacizumab
Started | 105
Completed | 70
Not Completed | 35
Not completed — Sponsor decision | 35

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 91
  Black or African American | 4
  Asian | 3
  American Indian or Alaska Native | 1
  Unknown | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate
Description: PFS rate at 18 months is defined as the percentage of participants who have not progressed or died within 18 months after niraparib combined with bevacizumab treatment initiation. Progression was assessed by response evaluation criteria in solid tumors (RECIST) version (v) 1.1 criteria per Investigator assessment and defined as a 20 percent (%) increase in the sum of the diameter of target lesions or unequivocal progression of existing non-target lesions. Survival rate is the percentage of participants without progression assessed by RECIST v1.1 or death by the landmark timepoint. Confidence intervals was constructed using exact method.
Time Frame: At 18 months
Population: Intent-to-treat (ITT) Population comprised of all participants who received any amount of niraparib (at least 1 dose).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Percentage of participants | 62 [51.9 to 71.2]

2. Secondary Outcome: Progression Free Survival (PFS) by RECIST v 1.1
Description: PFS was defined as the time from treatment initiation with niraparib combined with bevacizumab to the earlier date of assessment of progression, as assessed by RECIST v1.1 criteria, based on Investigator assessment, or death by any cause in the absence of progression.
Time Frame: Up to end of study (approximately 79 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Months | 19.6 [16.56 to 25.07]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the date of initiation of niraparib treatment in combination with bevacizumab to the date of death by any cause.
Time Frame: Up to end of study (approximately 79 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Months | 61.1 [44.88 to NA] — The upper limit of the 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events

4. Secondary Outcome: RECIST or Cancer Antigen (CA)-125 Progression Free Survival
Description: RECIST or CA-125 progression-free survival is defined as the time from initiation of niraparib treatment in combination with bevacizumab to the earliest date of progression assessed by RECIST v1.1 or CA-125 progression or death by any cause. CA-125 progression is defined as participants with elevated CA-125 pretreatment and normalization of CA-125 that must show evidence of CA-125 ≥ 2 × upper limit of normal (ULN) on 2 occasions at least 1 week apart OR elevated CA-125 pretreatment that never normalizes and must show evidence of CA-125 ≥ 2 × the nadir value on 2 occasions at least 1 week apart OR elevated CA-125 in the normal range pretreatment that must show evidence of CA-125 ≥ 2 × ULN on 2 occasions at least 1 week apart.
Time Frame: Up to end of study (approximately 79 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Months | 16.9 [13.27 to 22.05]

5. Secondary Outcome: Change From Baseline (CFB) in Functional Assessment of Cancer Therapy - Ovarian Symptom Index (FOSI)
Description: FOSI is a validated, 8-item measure of symptom response to treatment for ovarian cancer. Participants responded to their symptom experience over the past 7 days using a 5-point Likert scale scored from "not at all" (0) to "very much" (4). FOSI score was calculated as sum of item scores multiplied by 8 divided by number of items answered. The FOSI score ranged from 0 (severely symptomatic) to 32 (asymptomatic). A higher score indicated a better quality of life (QoL). Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1), Cycles 3, 5, 7, 9, 13, 17, 21, 25, 29 (Each Cycle was of 21 days) and end of treatment (70 months)
Population: ITT Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Scores on scale
  Baseline (Day 1) | 25.7 (3.79)
  CFB to Cycle 3: number analyzed (Participants) | 91
  CFB to Cycle 3 | -1.4 (4.30)
  CFB to Cycle 5: number analyzed (Participants) | 77
  CFB to Cycle 5 | -1.7 (3.89)
  CFB to Cycle 7: number analyzed (Participants) | 74
  CFB to Cycle 7 | -0.3 (3.09)
  CFB to Cycle 9: number analyzed (Participants) | 70
  CFB to Cycle 9 | -1.1 (3.74)
  CFB to Cycle 13: number analyzed (Participants) | 60
  CFB to Cycle 13 | -1.1 (4.25)
  CFB to Cycle 17: number analyzed (Participants) | 53
  CFB to Cycle 17 | -0.7 (3.39)
  CFB to Cycle 21: number analyzed (Participants) | 46
  CFB to Cycle 21 | -0.6 (3.77)
  CFB to Cycle 25: number analyzed (Participants) | 40
  CFB to Cycle 25 | 0.1 (3.73)
  CFB to Cycle 29: number analyzed (Participants) | 32
  CFB to Cycle 29 | 0.7 (3.40)
  CFB to End of Treatment (70 months): number analyzed (Participants) | 76
  CFB to End of Treatment (70 months) | -2.0 (5.21)

6. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: TFST was defined as the date of initiation of niraparib treatment in combination with bevacizumab treatment in the current study to the start date of the first subsequent anticancer therapy.
Time Frame: Up to end of study (approximately 79 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Months | 17.5 [14.55 to 20.73]

7. Secondary Outcome: Time to Second Subsequent Therapy (TSST)
Description: TSST was defined as the date of initiation of treatment of niraparib in combination with bevacizumab treatment in the current study to the start date of the second subsequent anticancer therapy.
Time Frame: Up to end of study (approximately 79 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Months | 38.6 [30.55 to 55.85]

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), Non-serious TEAEs and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. TEAEs is any AE that occurred for the first time after at least 1 dose of study treatment administration and until treatment duration. TEAEs which were not serious were considered as non-serious TEAEs. TESAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system. Percentages are rounded off to the nearest decimal point.
Time Frame: Up to end of treatment (70 months)
Population: Safety Population included all participants who received any amount of study treatment (i.e. any amount of bevacizumab or niraparib during the study).
Measure: Number; unit: Percentage of participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Percentage of participants
  TEAEs | 100
  Non-serious TEAEs | 100
  TESAEs | 30.5

9. Secondary Outcome: Number of Participants With TEAEs Leading to Niraparib Treatment Discontinuation
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. TEAE is any AE that occurred for the first time after at least 1 dose of study treatment administration. AEs were coded using the MedDRA coding system.
Time Frame: Up to end of treatment (70 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Participants | 46

10. Secondary Outcome: Number of Participants With TEAEs Leading to Niraparib Dose Reductions
Description: as for outcome 9
Time Frame: Up to end of treatment (70 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Participants | 81

11. Secondary Outcome: Number of Participants With AEs of Special Interest (AESI)
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs of scientific and medical concern related to the treatment were monitored, and rapidly communicated by investigator to sponsor. AEs were coded using the MedDRA coding system.
Time Frame: Up to end of treatment (70 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Participants
  New malignancies other than Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML) | 4
  MDS/AML Event | 2

12. Secondary Outcome: Change From Baseline (CFB) in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressures (DBP and SBP) were measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Millimeter of mercury (mmHg)
  SBP: Baseline (Day 1) | 129.7 (15.87)
  SBP: CFB to End of Treatment (70 months): number analyzed (Participants) | 96
  SBP: CFB to End of Treatment (70 months) | 2.8 (21.70)
  DBP: Baseline (Day 1) | 78.2 (9.30)
  DBP: CFB to End of Treatment (70 months): number analyzed (Participants) | 96
  DBP: CFB to End of Treatment (70 months) | 0.3 (11.17)

13. Secondary Outcome: Change From Baseline (CFB) in Pulse Rate
Description: Pulse Rate was measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Beats/minute
  Baseline (Day 1) | 80.6 (11.40)
  CFB to End of Treatment (70 months): number analyzed (Participants) | 95
  CFB to End of Treatment (70 months) | 4.3 (13.12)

14. Secondary Outcome: Change From Baseline (CFB) in Temperature
Description: Temperature was measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Celsius
  Baseline (Day 1) | 36.59 (0.297)
  CFB to End of Treatment (70 months): number analyzed (Participants) | 92
  CFB to End of Treatment (70 months) | -0.01 (0.439)

15. Secondary Outcome: Number of Participants Who Used Concomitant Medications
Description: Any permitted concomitant medication(s), including non-prescription medication(s) and herbal product(s), taken during the study were recorded.
Time Frame: Up to end of treatment (70 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Participants | 100

16. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameters: Basophils, Eosinophil, Leukocytes, Platelets, Lymphocytes, Monocytes and Neutrophils
Description: Blood samples were collected for the assessment of change from Baseline in hematology parameters. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Giga cells per liter (10^9 cells/L)
  Basophils: Baseline (Day 1): number analyzed (Participants) | 96
  Basophils: Baseline (Day 1) | 0.025 (0.0320)
  Basophils: CFB to End of Treatment (70 months): number analyzed (Participants) | 85
  Basophils: CFB to End of Treatment (70 months) | 0.008 (0.0385)
  Eosinophil: Baseline (Day 1): number analyzed (Participants) | 96
  Eosinophil: Baseline (Day 1) | 0.168 (0.3071)
  Eosinophil: CFB to End of Treatment (70 months): number analyzed (Participants) | 85
  Eosinophil: CFB to End of Treatment (70 months) | -0.028 (0.3245)
  Leukocytes: Baseline (Day 1) | 5.523 (1.5398)
  Leukocytes: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Leukocytes: CFB to End of Treatment (70 months) | 0.660 (3.9571)
  Platelets: Baseline (Day 1) | 219.810 (79.5186)
  Platelets: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Platelets: CFB to End of Treatment (70 months) | -6.585 (74.0943)
  Lymphocytes: Baseline (Day 1): number analyzed (Participants) | 102
  Lymphocytes: Baseline (Day 1) | 1.694 (0.6216)
  Lymphocytes: CFB to End of Treatment (70 months): number analyzed (Participants) | 91
  Lymphocytes: CFB to End of Treatment (70 months) | 0.152 (2.1904)
  Monocytes: Baseline (Day 1): number analyzed (Participants) | 102
  Monocytes: Baseline (Day 1) | 0.492 (0.2137)
  Monocytes: CFB to End of Treatment (70 months): number analyzed (Participants) | 91
  Monocytes: CFB to End of Treatment (70 months) | 0.007 (0.1819)
  Neutrophils: Baseline (Day 1): number analyzed (Participants) | 103
  Neutrophils: Baseline (Day 1) | 3.135 (1.1369)
  Neutrophils: CFB to End of Treatment (70 months): number analyzed (Participants) | 92
  Neutrophils: CFB to End of Treatment (70 months) | 0.197 (1.6063)

17. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter: Hemoglobin (Hb)
Description: Blood samples were collected for the assessment of change from Baseline in hematology parameter. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Grams per liter (g/L)
  Baseline (Day 1) | 116.800 (10.0234)
  CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  CFB to End of Treatment (70 months) | 4.787 (14.4303)

18. Secondary Outcome: Change From Baseline (CFB) in Hematology Parameter: Erythrocyte Mean Corpuscular Volume (MCV)
Description: as for outcome 17
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Femtoliters (fL)
  Baseline (Day 1) | 97.560 (7.0779)
  CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  CFB to End of Treatment (70 months) | 0.093 (5.4536)

19. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters: Urea Nitrogen, Glucose, Calcium, Chloride, Sodium, Magnesium and Potassium
Description: Blood samples were collected for the assessment of change from Baseline in clinical chemistry parameters. Baseline (Day 1) is defined as the most recent measurement prior to the first administration of study drug (including Cycle 1 Day 1).
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Millimoles per liter (mmol/L)
  Urea Nitrogen: Baseline (Day 1) | 5.681 (1.7222)
  Urea Nitrogen: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Urea Nitrogen: CFB to End of Treatment (70 months) | 0.375 (2.1948)
  Glucose: Baseline (Day 1) | 5.996 (2.3156)
  Glucose: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Glucose: CFB to End of Treatment (70 months) | -0.073 (2.8001)
  Calcium: Baseline (Day 1) | 2.377 (0.0872)
  Calcium: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Calcium: CFB to End of Treatment (70 months) | 0.018 (0.1005)
  Chloride: Baseline (Day 1) | 102.747 (2.9885)
  Chloride: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Chloride: CFB to End of Treatment (70 months) | -0.536 (3.4272)
  Sodium: Baseline (Day 1) | 139.467 (2.8184)
  Sodium: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Sodium: CFB to End of Treatment (70 months) | -0.298 (2.7192)
  Magnesium: Baseline (Day 1): number analyzed (Participants) | 102
  Magnesium: Baseline (Day 1) | 0.764 (0.1024)
  Magnesium: CFB to End of Treatment (70 months): number analyzed (Participants) | 86
  Magnesium: CFB to End of Treatment (70 months) | 0.017 (0.0977)
  Potassium: Baseline (Day 1) | 4.206 (0.3860)
  Potassium: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Potassium: CFB to End of Treatment (70 months) | 0.031 (0.4891)

20. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters: Bilirubin and Creatinine
Description: as for outcome 19
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Micromoles per liter (umol/L)
  Bilirubin: Baseline (Day 1) | 6.242 (2.8546)
  Bilirubin: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Bilirubin: CFB to End of Treatment (70 months) | 1.168 (3.2660)
  Creatinine: Baseline (Day 1) | 65.577 (16.3865)
  Creatinine: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Creatinine: CFB to End of Treatment (70 months) | 9.339 (16.4405)

21. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters: Albumin and Protein
Description: as for outcome 19
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
Grams per liter (g/L)
  Albumin: Baseline (Day 1) | 41.629 (3.3748)
  Albumin: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Albumin: CFB to End of Treatment (70 months) | 0.926 (3.1902)
  Protein: Baseline (Day 1) | 70.619 (5.0676)
  Protein: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  Protein: CFB to End of Treatment (70 months) | 0.309 (4.5744)

22. Secondary Outcome: Change From Baseline (CFB) in Clinical Chemistry Parameters: Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT)
Description: as for outcome 19
Time Frame: Baseline (Day 1) and end of treatment (70 months)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | Niraparib + Bevacizumab
Number analyzed (Participants) | 105
International units per Liter (IU/L)
  AST: Baseline (Day 1) | 24.619 (12.0043)
  AST: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  AST: CFB to End of Treatment (70 months) | 5.117 (20.0863)
  ALT: Baseline (Day 1) | 23.590 (13.4241)
  ALT: CFB to End of Treatment (70 months): number analyzed (Participants) | 94
  ALT: CFB to End of Treatment (70 months) | 4.362 (19.3484)

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected up to approximately 79 months (end of study) and treatment emergent non-serious adverse events and serious adverse events were collected up to 70 months (end of treatment).
Description: Safety Population included all participants who received any amount of study treatment (i.e. any amount of bevacizumab or niraparib during the study). All-cause mortality was reported for all enrolled participants
Arm/Group | Niraparib + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 56/105
Serious Adverse Events (participants affected / at risk) | 32/105
Other Adverse Events (participants affected / at risk) | 105/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib + Bevacizumab (N=105)
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 8
Small intestinal obstruction (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cystocele (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib + Bevacizumab (N=105)
Nausea (Gastrointestinal disorders) | 65
Constipation (Gastrointestinal disorders) | 40
Abdominal pain (Gastrointestinal disorders) | 34
Vomiting (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 31
Stomatitis (Gastrointestinal disorders) | 20
Abdominal distension (Gastrointestinal disorders) | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 72
Oedema peripheral (General disorders) | 16
Asthenia (General disorders) | 10
Chills (General disorders) | 6
Pain (General disorders) | 6
Pyrexia (General disorders) | 6
Headache (Nervous system disorders) | 59
Dizziness (Nervous system disorders) | 31
Neuropathy peripheral (Nervous system disorders) | 14
Peripheral sensory neuropathy (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 36
Neutropenia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 7
Platelet count decreased (Investigations) | 42
White blood cell count decreased (Investigations) | 23
Neutrophil count decreased (Investigations) | 18
Activated partial thromboplastin time prolonged (Investigations) | 14
Blood creatinine increased (Investigations) | 11
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 9
Weight increased (Investigations) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 38
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
Urinary tract infection (Infections and infestations) | 29
Upper respiratory tract infection (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 8
Hypertension (Vascular disorders) | 57
Hot flush (Vascular disorders) | 15
Proteinuria (Renal and urinary disorders) | 43
Haematuria (Renal and urinary disorders) | 9
Pollakiuria (Renal and urinary disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hyponatraemia (Metabolism and nutrition disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Insomnia (Psychiatric disorders) | 22
Anxiety (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 10
Palpitations (Cardiac disorders) | 12
Tachycardia (Cardiac disorders) | 10
Contusion (Injury, poisoning and procedural complications) | 9
Fall (Injury, poisoning and procedural complications) | 7
Pelvic pain (Reproductive system and breast disorders) | 6
Vision blurred (Eye disorders) | 8
Tinnitus (Ear and labyrinth disorders) | 6
Immune system disorders (Immune system disorders) | 11
Endocrine disorders (Endocrine disorders) | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Mouth ulceration (Gastrointestinal disorders) | 7
Blood alkaline phosphatase increased (Investigations) | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03326193/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT03326193/SAP_003.pdf